CLINICAL TRIAL: NCT04877366
Title: A Randomized, Double-blind, Placebo- and Active-Controlled, Single-Center, Three-time-period, Crossover Study to Evaluate the Effects of Sprinkled Format REDUCOSE on Post-Prandial Glycemic Response in Asian Patients with Type 2 Diabetes
Brief Title: Evaluate Effects of Sprinkled Format REDUCOSE in a Carbohydrate-rich, Mixed Meal on Post-prandial Glycemia
Acronym: Stardust
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2019CLI
Record Dates: First submitted 2021-04-28; First posted 2021-05-07 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Dietary Supplement

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ARM A: Sprinkled Format REDUCOSE (Active Comparator): 2 G powder sprinkle containing 250 mg REDUCOSE (mulberry leaf extract - 250 mg - 5% DNJ) + fiber, vitamin D, and chromium picolinate
  Interventions: Dietary Supplement: Dietary Supplement: Sprinkled Format REDUCOSE.
- ARM B: Placebo B: Standard Meal (Placebo Comparator): A placebo matching to the test product will be used as control
  Interventions: Other: Reference control
- ARM C: Placebo C: Acarbose (Placebo Comparator): Acarbose 100 mg tablet (provided in open-label format)
  Interventions: Other: Active comparator

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Sprinkled Format REDUCOSE. — 2 G powder sprinkle containing 250 mg REDUCOSE (mulberry leaf extract - 250 mg - 5% DNJ) + fiber, vitamin D, and chromium picolinate
  Arms: ARM A: Sprinkled Format REDUCOSE
Other: Reference control — A placebo matching to the test product will be used as control
  Arms: ARM B: Placebo B: Standard Meal
Other: Active comparator — Acarbose 100 mg tablet (provided in open-label format)
  Arms: ARM C: Placebo C: Acarbose

SUMMARY:
This is a mechanistic, single-center, double-blind, placebo- and active-controlled, three-time-period, crossover study to evaluate the effect of sprinkled format REDUCOSE compared to placebo (double-blind; confirmative) and active control (open-label; acarbose - explorative) on post prandial glycemia in Asian patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign written informed consent prior to study entry.
* Participants who self-identify as Asian; male or female, >18 years of age.
* Established diagnosis of type 2 diabetes (documented by either HbA1c 6.5 - 10.0% or a documented diagnosis of type 2 diabetes).
* Treatment naïve or on active therapy with metformin at a daily dose of 500-3000 mg at screening. Dose of metformin must have been stable for at least 3 months prior to screening.
* Participants must have a hematocrit value greater than or equal to 34.0% for females and 40% for males.
* Participants must have a hemoglobin value greater than or equal to 11.0 g/dL for females and 13.5 g/dL for males.

Exclusion Criteria:

* Fasting plasma glucose >220 mg/dl at screening.
* Impaired kidney function, eGFR of <60 mL/min/1.73 m2 at screening.
* BMI >35 kg/m2.
* Weight ≤ 50 kg.
* Elevated liver transaminase > 3 ULN at screening.
* Ongoing or recent (i.e. < 3 month) treatment with any oral or injectable glucose-lowering drug other than metformin.
* Ongoing or recent (i.e. < 3 month) injectable insulin therapy.
* Ongoing or recent (i.e. < 3 month) weight loss interventions (e.g. dietary weight loss programs) or any history of bariatric surgery or any documented weight loss >5% within previous 6 months.
* Ongoing or recent (i.e. < 3 month) treatment with anorectic drugs, systemic steroids, medications known to affect gastric motility, or any condition known to affect gastro-intestinal integrity and food absorption.
* Major medical/surgical event requiring hospitalization in the last 3 months.
* Known allergy and intolerance to product components or paracetamol.
* Alcohol intake higher than 2 servings per day. A serving is 0.4 dl of strong alcohols, 1 dl of red or white wine, or 3 dl of beer.
* Are unable to comply with protocol procedures in the opinion of the investigator.
* Have a hierarchical link with the research team members.
* Positive pregnancy test or breast-feeding at screening.
* Participants who have been dosed in another clinical study with any investigational drug/new chemical entity within 30 days or 5 half-lives (whichever is longer) prior to screening.
* Donation of blood or significant amount of blood loss within 8 weeks prior to screening. Participants must also agree to not donate blood within 8 weeks after their last visit.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Post-prandial glycemic excursion (ARMs A and B) | 0 ,15, 30, 60, 120, and 180 minutes.
  Incremental area under the curve post-prandial glycemic excursion (iAUC 0-1h, iAUC 0-2h, iAUC 0-3h).

SECONDARY OUTCOMES:
2h post-prandial glucose levels (ARMs A and B) | 0 ,15, 30, 60, and 120 minutes.
  Incremental area under the curve 2h post-prandial glucose levels
Total glucose (All ARMS) | 0 ,15, 30, 60, 120, and 180 minutes.
  Total glucose AUC 0-1h (tAUC 0-1h, tAUC 0-2h, tAUC 0-3h)
Plasma glucose iCmax (ARMs A and B) | 0 ,15, 30, 60, 120, and 180 minutes.
  Plasma glucose iCmax
Plasma glucose Tmax (ARMs A and B) | 0 ,15, 30, 60, 120, and 180 minutes.
  Plasma glucose Tmax
Plasma glucose AUC (ARMs A and B) | 0 ,15, 30, 60, 120, and 180 minutes.
  protocol states (iAUC 0-3h, tAUC 0-3h)
Serum insulin (All ARMs) | 0 ,15, 30, 60, 120, and 180 minutes.
  Serum insulin (iAUC 0-3h, iCmax, Tmax, tAUC 0-3h)
Plasma GLP-1 (ARMs A and B) | 0 ,15, 30, 60, 120, and 180 minutes.
  Plasma GLP-1 (iAUC 0-2h, iCmax, Tmax, tAUC 0-2h)
Plasma GIP (ARMs A and B) | 0 ,15, 30, 60, 120, and 180 minutes.
  Plasma GIP (iAUC 0-2h, iCmax, Tmax, tAUC 0-2h)
Plasma interleukin-6 (ARMs A and B) | 0 ,15, 30, 60, 120, and 180 minutes.
  Plasma interleukin-6 (IL-6) (iAUC 0-2h, iCmax, Tmax, tAUC 0-2h)
Gastric emptying (ARMs A and B) | 0 ,15, 30, 60, 120, and 180 minutes.
  Gastric emptying (iAUC 0-1h, tAUC 0-1h, iAUC 0-3h, tAUC 0-3h, Cmax and Tmax for paracetamol)
Matsuda Index (ARMs A and B) | 0, 30, 60, and 120 minutes.
  Matsuda Index

OTHER OUTCOMES:
Plasma glucose timepoints (ARMs A and B) | 0 ,15, 30, 60, 120, and 180 minutes.
  Plasma glucose at individual timepoints
Serum insulin timepoints (ARMs A and B) | 0 ,15, 30, 60, 120, and 180 minutes.
  Serum insulin at individual timepoints
Plasma GIP and GLP-1 (ARMs A and B) | 0 ,15, 30, 60, 120, and 180 minutes.
  Plasma GIP and GLP-1 at individual timepoints
Plasma IL-6 (ARMs A and B) | 0 ,15, 30, 60, 120, and 180 minutes.
  Plasma IL-6 at individual timepoints
Plasma GLP-1 iAUC (ARMs A and B) | 0 ,15, 30, 60, 120, and 180 minutes.
  Plasma GLP-1 (iAUC 0-1h, tAUC 0-1h)
Plasma GIP iAUC (ARMs A and B) | 0 ,15, 30, 60, 120, and 180 minutes.
  Plasma GIP (iAUC 0-1h, tAUC 0-1h)
Plasma IL-6 iAUC (ARMs A and B) | 0 ,15, 30, 60, 120, and 180 minutes.
  Plasma IL-6 (iAUC 0-4h, tAUC 0-4h, iAUC 0-2h, tAUC 0-2h, iAUC 0-1h, tAUC 0-1h)

CONTACTS AND LOCATIONS:
Locations (2):
- Orange County Research Center, Tustin, California, United States
- Temasek Polytechnic, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohamed M, Zagury RL, Bhaskaran K, Neutel J, Mohd Yusof BN, Mooney L, Yeo L, Kirwan BA, Aprikian O, von Eynatten M, Johansen OE. A Randomized, Placebo-Controlled Crossover Study to Evaluate Postprandial Glucometabolic Effects of Mulberry Leaf Extract, Vitamin D, Chromium, and Fiber in People with Type 2 Diabetes. Diabetes Ther. 2023 Apr;14(4):749-766. doi: 10.1007/s13300-023-01379-4. Epub 2023 Mar 1. PMID 36855010